CLINICAL TRIAL: NCT01986764
Title: Predictors of Healthy Mood and Memory After Oophorectomy
Brief Title: E2 and LDX for the Treatment of Cognitive Complaints After Oophorectomy
Acronym: E2LDX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not obtained for this study and no participants were enrolled.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, C. Neill Epperson, Associate Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 817642
Record Dates: First submitted 2013-10-30; First posted 2013-11-18 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Planned RRSO
Keywords: oophorectomy; RRSO; menopause; early menopause; cognition; memory; brain-imaging
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Lisdexamfetamine Dimesylate; Estradiol; Estrogens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- lisdexamfetamine (Active Comparator): lisdexamfetamine 20 mg/d to 60 mg/d for 12 weeks
  Interventions: Drug: Lisdexamfetamine
- Estradiol (Active Comparator): Estradiol 1 mg/d to 3 mg/d for 12 weeks
  Interventions: Drug: Estradiol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine
  Other Names: Vyvanse
  Arms: lisdexamfetamine
Drug: Estradiol
  Other Names: Estrogen
  Arms: Estradiol
Drug: Placebo — Placebo capsules will be filled with lactose powder.
  Arms: Placebo

SUMMARY:
This project seeks to address cognitive disturbance, which is a frequent adverse sequelae of riskreducing bilateral salpingo-oophorectomy (RRSO) with or without post-procedure chemotherapy and adjunctive treatments. RRSO after completion of childbearing is recommended for prevention of ovarian and breast cancer in women with BRCA1/BRCA2 mutations and standard of care for women with some forms of hormone-responsive cancer. Knowledge regarding the impact of this procedure, with or without chemotherapy, and subsequent hypogonadism on brain health is less than adequate. Premenopausal women who undergo an acute surgical menopause are at greater risk for verbal memory decline and executive function (EF) complaints, but as of yet, we cannot predict who is going to experience these adverse sequelae, nor do we have targeted prevention or treatment strategies other than hormone therapy, which is not an option in many cases and not always effective. An idealized sample as women who are planning for a RRSO will undergo brain imaging and behavioral assessments pre- and post-surgery as well as pre-/post-treatment with E2 or the psychostimulant, lisdexamphetamine (LDX; Vyvanse®).

ELIGIBILITY:
Inclusion Criteria:

Women ages 30 to 48 will be eligible for this study if they:

1. Have no previous or present history of a DSM-IV psychiatric disorder within the previous year or substance dependence disorder within the previous 5 years (psychostimulant abuse lifetime history), according to the Structured Clinical Interview for Diagnosis- DSM-IV (SCID)-Non-Patient Version;
2. Planning to undergo an oophorectomy or full hysterectomy;
3. Are premenopaual (have a baseline follicle stimulating hormone level (FSH) of <20 IU/ml);
4. Smoke < 10 cigarettes per day
5. Are right-handed;
6. Can provide proof of having had a gynecological exam and PAP test done within the previous 3 years at the time of screening;
7. Can provide proof of having had a mammogram within the previous 12 months at the time of screening;
8. Are able to give written informed consent;
9. Must have clear urine toxicology screen upon recruitment;
10. Are fluent in written and spoken English;
11. Negative urine pregnancy test.

Exclusion Criteria:

1. Mini-mental status exam score of less than or equal to 24;
2. Presence of a psychiatric disorder within previous year or a life time history of ADHD or psychotic disorder including bipolar disorder, schizoaffective disorder and schizophrenia;
3. Lifetime history of drug addiction or abuse, excepting nicotine;
4. Regular use of other psychotropic medication;
5. Regular use (more than once a week) of alcohol that is greater than 3 drinks per day;
6. Presence of a contraindication to treatment with stimulant medication; this would include the presence of hypertension (controlled or uncontrolled), coronary disease, atrial fibrillation, and arrhythmia;
7. History of seizures;
8. Presence of a contraindication to treatment with estrogen; this would include the presence of a history of blood clots, and estrogen-receptor positive breast cancer;
9. Claustrophobia;
10. History of cardiac disease including known cardiac defect or conduction abnormality;
11. Abnormal electrocardiogram during screening;
12. Current pregnancy or planning to become pregnant;
13. Presence of a metallic implant

Ages: 30 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
BADDS Score | 12 weeks
  This study uses a double-blind, placebo-controlled, design. The primary subjective outcome variable is the BADDS score measured at the initial screening visit, and one week after oophorectomy and 12 weeks after randomization to E2, LDX or placebo post-oophorectomy. The primary, out-of-scan objective outcome will be performance on the HVLT, while the primary, in-scanner outcomes will be behavioral and brain activation measures during performance of the N-back task.

SECONDARY OUTCOMES:
Cognitive Functioning | 12 weeks
  The secondary outcome variable studies changes in memory assessed using a battery of cognitive tasks.

CONTACTS AND LOCATIONS:
Overall Officials: C. Neill Epperson, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania, United States